CLINICAL TRIAL: NCT00741585
Title: Prognostic Value of the Circadian Pattern of Ambulatory Blood Pressure for Multiple Risk Assessment
Acronym: HYGIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Servicio Gallego de Salud (Other Government)
Responsible Party: Principal Investigator, Ramon C. Hermida, Professor, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYGIA; Hygia-2007-440
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Essential Hypertension; Cardiovascular Disease; Stroke; Chronic Kidney Disease
Keywords: Ambulatory blood pressure monitoring; Chronotherapy; Circadian; Non-dipper; Type 2 diabetes; Resistant hypertension; Total mortality
MeSH Terms: conditions — Essential Hypertension; Cardiovascular Diseases; Stroke; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — olmesartan; Irbesartan; candesartan; Telmisartan; Valsartan; Atenolol; Carvedilol; Doxazosin; lercanidipine; manidipine; Amlodipine; Ramipril; Enalapril; Lisinopril; Quinapril; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment with all prescribed hypertension medications on awakening
  Interventions: Drug: Any antihypertensive medication alone or in combination; Device: Ambulatory blood pressure monitoring
- 2 (Active Comparator): Treatment with at least one prescribed hypertension medication at bedtime
  Interventions: Drug: Any antihypertensive medication alone or in combination; Device: Ambulatory blood pressure monitoring

INTERVENTIONS:
Drug: Any antihypertensive medication alone or in combination — All drugs on awakening
  Other Names: Olmesartan; Irbesartan; Candesartan; Telmisartan; Valsartan; Atenolol; Carvedilol; Nevibolol; Doxazosine; Lercanidipine; Manidipine; Amlodipine; Ramipril; Enalapril; Lisinopril; Quinapril
  Arms: 1
Drug: Any antihypertensive medication alone or in combination — One or more drugs at bedtime
  Other Names: Olmesartan; Irbesartan; Candesartan; Telmisartan; Valsartan; Atenolol; Carvedilol; Nevibolol; Doxazosine; Lercanidipine; Manidipine; Amlodipine; Ramipril; Enalapril; Lisinopril; Quinapril
  Arms: 2
Device: Ambulatory blood pressure monitoring — Sampling at 20-min intervals from 07:00 to 23:00 and at 30-min intervals at night for 48 consecutive hours
  Other Names: ABPM

SUMMARY:
The HYGIA study was designed to investigate prospectively

1. the prognostic value of ambulatory blood pressure (BP) monitoring among subjects primarily evaluated at primary care settings
2. the impact of changes in ambulatory BP during follow-up in cardiovascular, cerebrovascular, metabolic, and renal risk in hypertensive patients
3. the influence of circadian time of treatment in cardiovascular, cerebrovascular, metabolic, and renal risk in hypertensive patients
4. the prevalence of an altered BP profile as a function of antihypertensive treatment, circadian time of treatment, age, and presence of diabetes, among other factors.

DETAILED DESCRIPTION:
Ambulatory blood pressure (BP) measurements (ABPM) correlate more closely with target organ damage and cardiovascular events than clinical cuff measurements. ABPM reveals the significant circadian variation in BP, which in most individuals presents a morning increase, small post-prandial decline, and more extensive lowering during nocturnal rest. However, under certain pathophysiological conditions, the nocturnal BP decline may be reduced (non-dipper pattern) or even reversed (riser pattern). This is clinically relevant since the non-dipper and riser circadian BP patterns constitute a risk factor for left ventricular hypertrophy, albuminuria, cerebrovascular disease, congestive heart failure, vascular dementia, and myocardial infarction. Hence, there is growing interest in how to best tailor and individualize the treatment of hypertension according to the specific circadian BP pattern of each patient.

The reduction of the normal 10-20% sleep-time BP decline that is characteristic of the non-dipper and riser patterns is indeed associated with elevated risk of target organ damage, particularly to the heart (left ventricular hypertrophy, congestive heart failure, and myocardial infarction), brain (stroke), and kidney (albuminuria and progression to end-stage renal failure). These results suggest that cardiovascular risk could be influenced not by BP elevation alone, but also by the magnitude of the circadian BP variability. However, the potential dimension of an altered BP profile is still under debate, as there is current discrepancy on the actual prevalence of a non-dipper BP profile among groups of interest, mainly the elderly, patients with diabetes and patients with resistant hypertension.

Moreover, several independent prospective studies have suggested that nighttime BP may be a better predictor of cardiovascular risk than daytime BP. Common to all previous trials is that prognostic significance of ABPM has relied on a single baseline profile from each participant, without accounting for possible changes in the BP pattern, mainly associated to antihypertensive therapy and aging during follow-up. Moreover, the potential benefit, i.e., reduction in cardiovascular risk, associated with the normalization of the circadian BP variability (e.g., conversion from non-dipper to dipper pattern) from appropriately envisioned treatment strategy is still a matter of debate.

The HYGIA study was designed to investigate, first, the comparative prognostic value of several BP parameters (including, among many others, BP variability, the diurnal/nocturnal ratio, diurnal and nocturnal means, hyperbaric index, slope of morning rise, etc) in the prediction of vascular, metabolic, and renal morbidity and mortality; second, whether potential changes in the circadian BP pattern after treatment with hypertension medications may be associated to changes in the risk of cardiovascular events, stroke, diabetes, and/or chronic kidney disease; and third, in keeping with the second major objective above, to further assess the potential changes in efficacy, safety profile, and/or capability of hypertension medications, used either alone or in combination, to modulate the circadian BP pattern and to reduce vascular, metabolic, and renal risks as a function of the circadian time of administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age.
* High-normal BP or essential hypertension.
* Any subject with recommendation for evaluation with ABPM according to the 2007 European Guidelines.
* Informed consent to participate in the study prior to any study procedures.

Exclusion Criteria:

* Known or suspected contraindications to any potential medication under investigation.
* Shift-workers.
* Inability to communicate and comply with all study requirements.
* Persons directly involved in the execution of this protocol.
* Intolerants to the use of the ABPM device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21983 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of circadian time of treatment in cardiovascular, cerebrovascular, metabolic, and renal risk assessment. | Yearly evaluation for at least ten years

SECONDARY OUTCOMES:
To evaluate the influence of circadian time of treatment in BP control of hypertensive patients. | Yearly evaluation for at least ten years
To evaluate the prevalence of an altered (non-dipper) BP profile in patients with resistant hypertension as a function of the circadian time of treatment. | Yearly evaluation for at least ten years
To evaluate the influence of diabetes and circadian time of treatment in the prevalence of an altered (non-dipper) BP profile. | Yearly evaluation for at least ten years
To evaluate the influence of age and circadian time of treatment in the prevalence of an altered (non-dipper) BP profile. | Yearly evaluation for at least ten years
To evaluate, for all groups of interest, the prevalence and vascular, metabolic, and renal risk profile of white-coat hypertension. | Yearly evaluation for at least ten years
To evaluate, for all groups of interest, the prevalence and vascular, metabolic, and renal risk profile of masked hypertension. | Yearly evaluation for at least ten years
To evaluate, for all previous objectives, potential differences between men and women. | Yearly evaluation for at least ten years
To evaluate the impact of changes in ambulatory BP in vascular, metabolic, and renal risk assessment. | Yearly evaluation for at least ten years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, PhD, Study Director — University of Vigo
Locations (20):
- Spain (20):
  - CS Friol, Friol, Lugo
  - CS A Estrada, A Estrada, Pontevedra
  - CS Baiona, Baiona, Pontevedra
  - CS Bueu, Bueu, Pontevedra
  - CS A Guarda, La Guardia, Pontevedra
  - CS Valmiñor, Nigrán, Pontevedra
  - CS Panxón, Nigrán, Pontevedra
  - CS Tomiño, Tomiño, Pontevedra
  - Bioengineering & Chronobilogy Labs., University of Vigo, Vigo, Pontevedra
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - CS Calle Cuba, Vigo, Pontevedra
  - CS A Doblada, Vigo, Pontevedra
  - CS Coia, Vigo, Pontevedra
  - CS Sardoma, Vigo, Pontevedra
  - CS Teis, Vigo, Pontevedra
  - CS Vilaboa, Vilaboa, Pontevedra
  - CS San Roque, Vilagarcía de Arousa, Pontevedra
  - CS Fingoi, Lugo
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - CS Lerez, Pontevedra

REFERENCES:
- [Derived] Hermida RC, Crespo JJ, Dominguez-Sardina M, Otero A, Moya A, Rios MT, Sineiro E, Castineira MC, Callejas PA, Pousa L, Salgado JL, Duran C, Sanchez JJ, Fernandez JR, Mojon A, Ayala DE; Hygia Project Investigators. Bedtime hypertension treatment improves cardiovascular risk reduction: the Hygia Chronotherapy Trial. Eur Heart J. 2020 Dec 21;41(48):4565-4576. doi: 10.1093/eurheartj/ehz754. PMID 31641769
- [Derived] Hermida RC. Sleep-time ambulatory blood pressure as a prognostic marker of vascular and other risks and therapeutic target for prevention by hypertension chronotherapy: Rationale and design of the Hygia Project. Chronobiol Int. 2016;33(7):906-36. doi: 10.1080/07420528.2016.1181078. Epub 2016 May 24. PMID 27221952